CLINICAL TRIAL: NCT07190014
Title: Investigation of the Effects of a Virtual Reality Application Developed for the Assessment of Cervical Joint Range of Motion and Joint Position Sense
Brief Title: Virtual Reality Application for Assessing Neck Movement and Position Sense
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assistant Professor of Neurological Physiotherapy and Rehabilitation, Hacettepe University
Other Study IDs: VRROMJPSEV
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neck Pain
Keywords: virtual reality; neck pain; pain; chronic pain; evaluation; range of motion; joint position sense; proprioception; application; technologic rehabilitation
MeSH Terms: conditions — Neck Pain; Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Virtual Reality Based Assesment Group - Participants with Chronic Neck Pain: Participants in this group will be evaluated with the virtual reality assessment module developed by our team.
  * Cervical range of motion (ROM): The module records movement angles in six directions - flexion, extension, right/left lateral flexion, and right/left rotation.
  * Joint position sense (JPS): For this assessment, participants move their head to 65% of their available range in a given direction, return to the neutral position, and then attempt to reposition to the same target. Errors are recorded in degrees.
  Results from the VR module will be compared with those obtained using the Cervical Range of Motion (CROM) device.
- CROM Based Assesment Group - Participants with Chronic Neck Pain: Participants in this group will be evaluated using the Cervical Range of Motion (CROM) device, a standard clinical tool for neck assessment.
  * Cervical range of motion (ROM): Movement angles will be measured in six directions - flexion, extension, right/left lateral flexion, and right/left rotation.
  * Joint position sense (JPS): Participants will be guided to move their head to 65% of the available range in a given direction, return to the neutral position, and then attempt to reposition to the same target. Errors will be recorded in degrees.
  Measurements obtained from the CROM device will be compared with those from the virtual reality assessment module.
- Virtual Reality Based Evaluation - Healthy Participiants: Participants in this group will be evaluated with the virtual reality assessment module developed by our team. • Cervical range of motion (ROM): The module records movement angles in six directions - flexion, extension, right/left lateral flexion, and right/left rotation. • Joint position sense (JPS): For this assessment, participants move their head to 65% of their available range in a given direction, return to the neutral position, and then attempt to reposition to the same target. Errors are recorded in degrees. Results from the VR module will be compared with those obtained using the Cervical Range of Motion (CROM) device.
- CROM Based Assesment Group - Healthy Participants: Participants in this group will be evaluated using the Cervical Range of Motion (CROM) device, a standard clinical tool for neck assessment. • Cervical range of motion (ROM): Movement angles will be measured in six directions - flexion, extension, right/left lateral flexion, and right/left rotation. • Joint position sense (JPS): Participants will be guided to move their head to 65% of the available range in a given direction, return to the neutral position, and then attempt to reposition to the same target. Errors will be recorded in degrees. Measurements obtained from the CROM device will be compared with those from the virtual reality assessment module.

SUMMARY:
The goal of this observational study is to examine whether a virtual reality application developed by our team can be used to evaluate cervical range of motion (ROM) and joint position sense (JPS) in individuals with chronic neck pain.

The main questions it aims to answer are:

* Does the virtual reality application provide reliable measurements of cervical ROM?
* Does the application accurately assess cervical JPS when compared with a standard clinical tool (Cervical Range of Motion device, CROM)?

Researchers will compare results from the VR application with results from the CROM device to see if the two methods give similar outcomes.

Participants will:

* Complete a demographic and clinical evaluation.
* Perform standardized neck movements (flexion, extension, left/right lateral flexion, left/right rotation).
* Be assessed using both the CROM device and the VR application for ROM and JPS.

DETAILED DESCRIPTION:
Neck pain is one of the most common musculoskeletal problems and is associated with limitations in mobility and proprioceptive deficits. Reliable assessment of cervical range of motion (ROM) and joint position sense (JPS) is critical for both clinical evaluation and rehabilitation planning. Traditional devices, such as the Cervical Range of Motion (CROM) instrument, are widely used but have limitations, including the need for manual operation, restricted visualization, and lower potential for patient engagement.

Virtual reality (VR) technologies provide an opportunity to overcome these limitations by offering objective measurements, immersive feedback, and greater standardization of the testing environment. Our team has developed a VR-based application specifically designed to assess cervical ROM and JPS. This application may contribute to more accurate, reliable, and user-friendly evaluation methods compared to conventional tools.

In this observational study, individuals with chronic neck pain will be assessed using both the CROM device and the VR application. The study will compare the results obtained from both methods to determine the validity and reliability of the VR-based system.

The findings are expected to provide evidence for the clinical use of VR in musculoskeletal assessment, potentially enhancing diagnostic accuracy and supporting the development of innovative rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Neck Pain (CNP) participants

  * Age 18-65. ￼
  * ≥ 6 months of neck pain. ￼
  * Willing to participate (informed consent). ￼

Healthy volunteers

* Age 18-65. ￼
* No neck pain complaints. ￼
* Willing to participate (informed consent). ￼

Exclusion Criteria:

* Prior adverse virtual reality experience. ￼

  * Photophobia: UPSIS-12 score > 12. ￼
  * Migraine screen: ≥2 "yes" on ID-Migraine. ￼
  * Any neurological deficit. ￼
  * History of spinal surgery. ￼
  * Medical conditions that could interfere with participation: orthopedic, inflammatory, cardiovascular, rheumatologic, or vestibular problems. ￼
  * Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from individuals referred to the Neurosurgery Department of Hacettepe University, Ankara, Türkiye, as well as healthy volunteers from the general population. The study population will include adults within the target age range, consisting of both individuals with chronic neck pain and healthy controls, to allow comparison between clinical and non-clinical groups.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion (ROM) Measurements | At baseline, during a single assessment session (Day 1).
  Cervical ROM will be assessed in six directions (flexion, extension, right/left lateral flexion, right/left rotation). Measurements will be obtained using both the CROM device and the virtual reality assessment module developed by the research team. Results will be compared to evaluate the validity of the VR-based system.
Cervical Joint Position Sense (JPS) Error | At baseline, during a single assessment session (Day 1).
  JPS will be evaluated by asking participants to move their head to 65% of the available ROM in a given direction, return to the neutral position, and then attempt to relocate the same target position. Errors will be recorded in degrees. Measurements will be taken with both the CROM device and the VR assessment module, and results will be compared.

SECONDARY OUTCOMES:
Usability and Participant Experience | Immediately after completion of the VR assessment session (Day 1).
  Participants' feedback on the ease of use, comfort, and overall experience of the virtual reality application will be collected using a structured questionnaire.
Simulator Sickness Questionnaire (SSQ) Scores | Immediately after completion of the VR assessment session (Day 1).
  Simulator Sickness Questionnaire (SSQ) Scores VR-related side effects, such as dizziness, nausea, or eye strain, will be assessed using the Simulator Sickness Questionnaire (SSQ), a 16-item self-report scale. Each symptom is rated from 0 (none) to 3 (severe), and weighted total scores range from 0 (no symptoms) to 235 (maximum symptoms). Higher scores indicate more severe simulator sickness symptoms (worse outcome).
Assessment Duration | During the single assessment session (Day 1).
  The total time required to complete the ROM and JPS evaluations will be recorded for both the VR application and the CROM device. This will allow comparison of the efficiency of the two assessment methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospital Department of Neurosurgery, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share individual participant data because of privacy and confidentiality concerns.

REFERENCES:
- [Background] Sarig Bahat H, Takasaki H, Chen X, Bet-Or Y, Treleaven J. Cervical kinematic training with and without interactive VR training for chronic neck pain - a randomized clinical trial. Man Ther. 2015 Feb;20(1):68-78. doi: 10.1016/j.math.2014.06.008. Epub 2014 Jul 5. PMID 25066503